CLINICAL TRIAL: NCT06129019
Title: Investigation of the Effect of Reiki Application on Depression, Anxiety and Physical Activity in Individuals Diagnosed With Relapsing-Remitting Multiple Sclerosis
Brief Title: the Effect of Reiki Application on Depression, Anxiety and Physical Activity in Patient With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22/11
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: reiki; anxiety; physical activity
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Anxiety Disorders; Motor Activity | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: (Experimental): Reiki application will be done
  Interventions: Behavioral: Reiki
- Control (No Intervention): Reiki application will not be done

INTERVENTIONS:
Behavioral: Reiki — Reiki application will be done
  Arms: Experimental:

SUMMARY:
During Reiki application, individuals may report feeling a slight warm sensation under and near the therapist's hand. The only rule in Reiki practice is that the individual must give permission to the practitioner to facilitate the flow of energy. The person receiving Reiki during the application does not have to believe in Reiki. Because Reiki is universal life energy and is available to everyone. Reiki is generally safe and no serious side effects have been reported. Reiki practice in the last 10 years; It is increasing among physicians, nurses and other healthcare professionals.

This study was planned to investigate the effect of reiki application on depression, anxiety and physical activity in individuals diagnosed with Relapsing-Remitting Multiple Sclerosis.

Geri bildirim gönder Yan paneller

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Having the ability to use technological devices
* Not using Reiki and similar integrative treatment methods
* No verbal communication disability (hearing and speaking)
* Not having a diagnosed psychiatric disorder
* Patients who have been receiving Relapsing-Remitting MS treatment for more than three months

Exclusion Criteria:

* Patients using any complementary alternative treatment methods
* Patients who cannot communicate by phone to participate in remote reiki application
* Patients with autoimmune diseases other than multiple sclerosis
* Patients with communication disabilities
* Patients with another known neurological system disease (dementia, Alzheimer's, etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Beck Depression Scale | 4 week
  The scale was administered to investigate each participant's feelings and attitudes regarding the general depressive state. Each patient was asked to read several groups of statements and then mark the one statement in each group that best described how he or she felt "during the past week." BDI, which evaluates four statements describing increasing intensities of depressive symptoms between 0 and 3 points, includes 21 items. Depressive symptoms were classified as follows: minimal-to-moderate depressive symptoms (range 14 to 19), moderate-to-severe depressive symptoms (range 20 to 29), severe depressive symptoms (range 30 to 63).
Beck Anxiety Scale | 4 week
  BAI is a self-rating scale developed by Beck et al. (1988) and used to determine the frequency of anxiety symptoms experienced by individuals. It is a Likert-type scale consisting of 21 items and scored between 0-3. Its validity and reliability in Turkey were determined by Ulusoy et al.
International Physical Activity Survey | 4 week
  There are some scales that can be used in primary care to evaluate physical mobility. One of these is the "International Physical Activity Questionnaire", which was developed by the International Consensus Group consisting of researchers from various countries with the support of the World Health Organization and the Center for Disease Control, to be used to measure physical activity and inactivity in 1997 and 1998; (IPAQ)" is a standard tool. Reliability and/or validity studies were conducted in 14 centers from 12 countries in 2000 for at least two of the four long (IPAQ-long) and four short (IPAQ-SF) forms of the IPAQ. This scale was adapted into Turkish as long form (UF) and short form (SF) under the name "International Physical Activity Questionnaire (UFAA)" and its validity and reliability study was conducted by Sağlam et al. in 2010

CONTACTS AND LOCATIONS:
Locations (1):
- Firat University, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No